CLINICAL TRIAL: NCT01471977
Title: Interventions to Promote Adherence to Tuberculosis Treatment Among Patients Attending Basic Medical Unit of Taluka Gambat, Pakistan
Brief Title: Treatment Adherence of Tuberculosis Medicines
Acronym: TBAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gambat Institute of Medical Sciences (Industry)
Responsible Party: Principal Investigator, Maliha Naseer, senior resident, Gambat Institute of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB
Record Dates: First submitted 2011-11-04; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Educational Status; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- education, counselling, default tracer (Experimental)
  Interventions: Other: education,counseling, default tracers,quality of care

INTERVENTIONS:
Other: education,counseling, default tracers,quality of care — these interventions were administered along with standard treatment i.e. DOTS at the time of standard follow up of patients at clinic
  Other Names: tuberculosis; directly observed short course treatment; education and counseling; default tracer

SUMMARY:
It was hypothesized that tuberculosis patients receiving multiple interventions like educations, counseling and default tracing along with DOTS were more likely to adhere to tuberculosis treatment as compared to few interventions or DOTS only.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* > 18years
* either sex
* diagnosed to have tuberculosis through chest x ray or sputum microscopy
* eligible to participate in the study

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients cured | 8 months
  Cured: If the patient was sputum smear positive (ss+ve) at the time of enrollment, completed treatment, Had negative smear on 2 occasions during follow-up
Proportion of patients completed treatment | 8 months
  Treatment completed: SS+ve, or SS-ve or extra-pulmonary, had a negative smear result at the end of intensive phase but no smear result at the end of treatment completed 8 month treatment
Proportion of patients died | 8 months
  died during the course of treatment
proportion of patients defaulted | 8 months
  not collected drugs for more than 2 consecutive months either sputum smear positive or negative
proportion of patients with treatment failure | 8 months
  Treatment failure: SS+ve, found to be smear positive at 5th month or later or SS-ve found to be smear positive at 2nd month
proportion of patients transferred out | 8 months
  Transferred to another TB register

CONTACTS AND LOCATIONS:
Overall Officials: Nisar Sheikh, MBBS, Principal Investigator — GIMS
Locations (1):
- Basic Medical Unit of Taluka Gambat, Khairpur, Sindh, Pakistan